CLINICAL TRIAL: NCT01800630
Title: An Open Label, Phase 1, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Clinical Activity of Gemcitabine Hydrochloride Oral Formulation(D07001-F4) in Patients With Advanced Solid Malignancies and Malignant Lymphomas
Brief Title: Phase1 Study of Gemcitabine HCl Oral Formulation(D07001-F4) in Patients With Advanced Solid Malignancies and Malignant Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InnoPharmax Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HR-12-001
Record Dates: First submitted 2013-02-23; First posted 2013-02-28 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Advanced Solid Malignancies; Malignant Lymphomas
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine HCl Oral Formulation (D07001-F4) (Experimental): Subjects will receive a single 5-mg (nontherapeutic) dose of gemcitabine (Gemzar®) via an IV push and then treated with Gemcitabine HCl Oral Formulation (D07001-F4)according to assigned cohort (2 mg to 80 mg) on Day 1, 3, 5, 8, 10, and 12 of 4 21-day cycles study treatment period.
  Interventions: Drug: Gemcitabine HCl Oral Formulation

INTERVENTIONS:
Drug: Gemcitabine HCl Oral Formulation
  Other Names: D07001-F4

SUMMARY:
Open-label Phase 1 sequential dose-escalation study of 10 increasing doses (3 to 6 patients each)to determine and characterize the DLTs and MTD of gemcitabine HCl oral formulation (D07001-F4). Patients will be assigned to receive oral D07001-F4 on Days 1, 3, 5, 8, 10, and 12 of 4 21-day cycles each to further characterize safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 20 years and older
* Signed and dated informed consent form
* Patients with advanced solid malignancies and malignant lymphomas with histological or pathologic confirmation who have failed standard therapies or for which no standard therapy exists
* Both measurable and non-measurable disease allowed (measurable disease per RECIST, version 1.1, or Revised Response Criteria for Malignant Lymphoma [Cheson criteria])
* World Health Organization (WHO) performance status 0 to 2
* At least 28 days have elapsed (before screening) since the patient's prior systemic therapy, radiotherapy, or any major surgery (excluding diagnostic biopsy or venous access device placement)
* Patient has

  * Absolute neutrophil count (ANC) ≥ 1500 cells/mm³
  * Platelet count ≥ 75,000 cells/mm³
  * Hemoglobin ≥ 9 g/dL.
* Patient has adequate liver function, demonstrated by:

  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5*the upper limit of normal (ULN) (≤ 5.0*ULN in case of liver metastasis)
  * Total bilirubin ≤ 1.5 mg/dL (unless due to Gilbert's syndrome)
  * Albumin ≥ 2.5 g/dL
  * International normalized ratio (INR) < 1.5
* Patient has adequate renal function:

  * Serum creatinine ≤ 1.5*ULN.
* Patient has a life expectancy > 12 weeks.
* If a woman of child-bearing potential, patient has a negative pregnancy test and is not breast feeding.
* If a woman of child-bearing potential, patient is using a medically acceptable form as two barrier methods (e.g., combination of condom, diaphragm, intrauterine device), hormonal contraception (estrogen or progesterone agents) or one barrier method in combination with spermicide. Birth control is required 1 month prior to screening, for the duration of their study participation, and for 1 month after the end of the study; female partners of male patients will also adhere to similar birth control methods
* Patient is willing to comply with protocol-required visit schedule and visit requirements

Exclusion Criteria:

* Patient is receiving full-dose (therapeutic) anticoagulation therapy.
* Patient is intolerant or allergic or has a known hypersensitivity to gemcitabine
* Patient has clinically significant cardiovascular disease (for example: uncontrolled hypertension, unstable angina, congestive heart failure, or New York Heart Association Grade 2 or greater).
* Patient has uncontrolled serious cardiac arrhythmia.
* Patient has known brain metastases or any leptomeningeal metastases.
* Patient has any unresolved toxicity (>Grade 1) from previous anticancer therapy with the exception of renal and liver function which are required to be in the range as described in inclusion criteria and peripheral neuropathy acceptable if resolved to at least grade 2.
* Patient has received radiotherapy of more than 10 Gy within 6 months of screening.
* Patient has a history of drug or alcohol abuse within last year.
* Patient has documented cerebrovascular disease.
* Patient has a seizure disorder not controlled on medication (based on decision of Investigator).
* Patient received an investigational agent within 28 days of screening
* Patient received systemic treatment for infection within 14 days of screening.
* Patient has known human immunodeficiency virus (HIV) infection.
* Patient has hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection in medical history.
* Patient has received yellow fever vaccine and other live attenuated vaccines within the last 4 weeks
* Patient has any other serious medical condition that, in the Investigator's medical opinion, would preclude safe participation in a clinical trial.
* Patients have gastrointestinal disease/prior surgery that may interfere with adequate oral therapy absorption
* Patients after allogeneic stem cell transplantation
* Patients with less than 12 months from autologous stem cell transplantation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-04; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To determine MTD and DLT of Gemcitabine Oral formulation | During the 21-day cycle 1 treatment
  MTD will be determined by study structure and DLT will be determined by definition

SECONDARY OUTCOMES:
AE/SAE incidences | Throughout treatment and 30-day follow-up (estimated average of 5 months)
  AEs will be assessed via the CTCAE version 4.03
Changes from baseline in clinical laboratory test (hematology, biochemistry, coagulation factors and urinalysis) results, vital sign measurements, physical examination findings, and ECG and 2D echocardiogram/multiple-gated acquisition (MUGA) scan results | Throughout treatment and 30-day follow-up (estimated average of 5 months)
characterize the PK of D07001-F4 | cycle 0 and cycle 1 (Day -7~Day 19)
ORR(Objective Response Rate) and tumor response | After cycle 2 and cycle 4 treatments (estimated average of 2 months and 4 months)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chi Lin, MD, Principal Investigator — National Taiwan University Hospital; Wu-Chou Su, MD, Principal Investigator — National Cheng-Kung University Hospital; Yee Chao, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (3):
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei